CLINICAL TRIAL: NCT04951089
Title: Comparison of the Clinical Performances of Air-Q SP 3G and i-Gel by Novice Intubators During Manual In-line Neck Stabilization: A Randomized Controlled Trial
Brief Title: Comparison of the Clinical Performances of Air-Q SP 3G and i-Gel
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS GAITINI MD, Associate Clinical Prpfessor of Anesthesiology, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0087-21-BNZ
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia
Keywords: Supraglottic devices; Airway; Insertion success

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-gel supraglottic device insertion for oxygenation (Experimental): i-gel supraglottic device insertion for oxygenation i-gel supraglottic device insertion for oxygenation and ventilation
  Interventions: Device: i-gel Supraglottic device insertion
- Air-Q SP 3G supraglottic insertion for oxygenation (Experimental): Air-Q SP 3G supraglottic device insertion for oxygenation Air-Q SP 3G supraglottic device insertion for oxygenation and ventilation
  Interventions: Device: Air-Q SP 3G Supraglottic device insertion

INTERVENTIONS:
Device: i-gel Supraglottic device insertion — i-gel insertion for oxygenation
  Arms: i-gel supraglottic device insertion for oxygenation
Device: Air-Q SP 3G Supraglottic device insertion — Air-Q SP 3G insertion for oxygenation
  Arms: Air-Q SP 3G supraglottic insertion for oxygenation

SUMMARY:
Establishing a definitive airway defined as a tube placed in the trachea with cuff inflated below the vocal cords is the first priority in the airway management of the pre-hospital trauma patient, according to the last edition of the Advanced Trauma Life Support (ATLS) textbook, of the American College of Surgeons. However, studies revealed that the success rate of tracheal intubation in the prehospital setting using direct laryngoscopy (DL), the standard intubation technique is suboptimal. The Advance Trauma Life Support suggested the use of Supraglottic Airway Devise (SAD) in managing the difficult airway. The air-Q SP 3G was introduced as an alternative for managing the difficult airway. The i-gel is proposed as supraglottic device made of a medical grade thermoplastic elastomer. The unique design of both devices is that a cuff is not needed to be inflated .

A randomize controlled trail will be conduce. Participants will insert the both supraglottic devices to compare performance of ventilation and oxygenation of the patients.

The insertion will be performed on age 18-75 year patients, scheduled for elective surgery with general anesthesia. The SAD use in the study will be a single use i-gel size 4 or 5 and the air-Q SP 3G- size 4 or 5 For induction of anesthesia all patients will receive premedication. After 3 min of preoxygenation anesthesia will induce with up to 2 mcg/Kg fentanyl and 2-3 mg propofol Neuromuscular blockade will be obtained with rocuronion.

The participant will performed one insertion of the i-gel or the air-Q SP 3G on the patient while manual in-line stabilization of the neck Primary outcome: time to success insertion of SAD Secondary outcome : duration in seconds of insertion

DETAILED DESCRIPTION:
In the combat setting, airway compromise is the second leading cause of preventable death after hemorrhage.

Establishing a definitive airway defined as a tube placed in the trachea with cuff inflated below the vocal cords is the first priority in the airway management of the pre-hospital trauma patient, according to the last edition of the Advanced Trauma Life Support (ATLS) textbook, of the American College of Surgeons. However, studies revealed that the success rate of tracheal intubation in the prehospital setting using direct laryngoscopy (DL), the standard intubation technique is suboptimal.

Possible reasons for the failure in achieving definitive airway in trauma patients are the requirement for in-line stabilization of the neck, and the inexperience of the providers.

The Tactical Combat Casualty Care (TCCC) Guidelines recommend using a supraglottic airway device (SAD) as an option to assist in securing the airway in tactical evacuation phase of care.

In a recent published Randomized Control Trail in patients, the success of blind intubation did not support the use of tracheal intubation (TI) via iLTS-D by novice intubators. However, this study revealed a high success rate (84.6%) of iLTS-D placement in the oropharynx, associated with effective ventilation as confirmed by capnography.

The time to obtain successful iLTS-D placement in the oropharynx was 42 sec, which is 2.5 times shorter than the time to achieve TI with DL.

These results encourage the use of a second generation Supraglottic Airway Device (SAD) by novice intubators as the first airway intervention in trauma patients, who require immediate airway management.

SADs play a key role as primary and rescue devices in predicted and unanticipated difficult airway management, by providing both a patent airway for oxygenation and ventilation and a conduit for TI, thereby avoiding the disastrous outcomes of 'cannot intubate, cannot oxygenate' situations.

Recently study reported the effectiveness of initial insertion with Laryngeal Tube (LT) vs initial Endotracheal Intubation (ETI) in adults out of Hospital cardiac arrest (OHCA).This study concludes that a strategy of initial LT insertion was associated with significantly greater 72-hour survival compare with the strategy of initial ETI.

These findings suggest that SAD insertion may be considered as an initial airway management strategy in patients with OHCA.

The implication of the SAD effectivity in fasting rescue the airway pattern and reassure oxygenation is greatest importance in combat setting.

The self-pressurized air-Q intubating laryngeal airway (air-Q SP 3G) (Mercury Medical, Clearwater, FL, USA) is a single-use SAD that does not require cuff inflation. The original air-Q intubating laryngeal airway (Cookgas LLC; Mercury Medical) was designed to facilitate tracheal intubation through its lumen.

The air-Q SP 3G differs from the original air-Q by the absence of an inflatable cuff and the continuity between the airway tube and cuff through an inner aperture at the junction the airway tube and periglottic cuff of the air-Q SP 3G makes the intracuff pressure equilibrate dynamically with the airway pressure and is designed to adjust to the patient's pharyngeal and periglottic anatomy .

The absence of a pilot balloon and continuity between the airway tube and the cuff through an inner aperture has several clinical benefits when compared with other cuffed SAD.

First, the provider does not loose time with the inflation cuff maneuver. Second, intra-cuff pressures are determined by the airway pressures, because of the equalization of pressures with the movement of gas between the cuff and airway tube.

Third, lower intra-cuff pressures are maintained overall as a result of being limited by the peak airway pressures, with the highest pressures exerted during inspiration. Fourth, by not exceeding peak airway pressures, the balance between intra-cuff pressures and the airway seal of the device may be optimized at lower pressure. Therefore, the risk of sore throat, neuropraxic injury, and gastric insufflation seen with overinflation of traditional cuffed supraglottic devices may be reduced.

Recently, the air-Q SP 3G has been upgraded with the addition of the gastric channel in order diminish the risk of aspiration.

The i-gel second generation SAD, disposable airway (Intersurgical Ltd, Workingham, UK) is a SAD made of a medical grade thermoplastic elastomer. Its unique design does not need an inflatable cuff because the thermoplastic elastomer provides the seal. The i-gel is gaining a reputation for its ease of insertion and for its use in many clinical situations. Previous studies have demonstrated that the i-gel can be placed more faster than conventional laryngeal mask airways, which might play a role in prehospital settings. Other advantages of the i-gel are ease of training, cost, safety, and simplicity of use.

There have been no studies comparing these devices in patients with limited neck extension. Therefore, the aim is to compare the clinical performance of these two devices in adult patients with simulated cervical immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Patient ASA ( American Society Anesthesiologist) I-II
* non pregnancy

Exclusion Criteria:

* Difficult airway
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Insertion success ratio between supraglottic device the i-gel and Air-Q SP 3G Comparison of the insertion success in the oropharynx of the i-gel and the Air-Q SP 3G supraglottic devices, insertion success detected by capnography trace | From insertion of supraglottic between the lips of the subject to final success or failure of insertion 30 seconds
  Comparison of the insertion success in the oropharynx of i-gel and the Air-Q SP 3G supraglottic devices, insertion success detected by capnography trace